CLINICAL TRIAL: NCT07068945
Title: Study of the Transition From Child Psychiatry to Adult Psychiatry in Nice Within a Population of 17-year-old Adolescents
Acronym: Odysee3
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 25-HPNCL-04 Odysee3
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Child Psychiatry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of 17-year-old patients living in Nice and receiving psychiatric care: Group of 17-year-old patients living in Nice and receiving psychiatric care
  Interventions: Behavioral: Group of 17-year-old patients living in Nice and receiving psychiatric care

INTERVENTIONS:
Behavioral: Group of 17-year-old patients living in Nice and receiving psychiatric care — Prospective study aiming to determine the annual prevalence of 17-year-old patients living in Nice who attend hospital-based child and adolescent psychiatry services. Secondary objectives include: estimating prevalence among under-18 psychiatric patients; describing clinical and sociodemographic profiles (sample of 100 patients); mapping 1-year care trajectories; evaluating clinical outcomes; assessing transition preparedness (to adult psychiatry); and identifying factors associated with psychiatric care continuity at 12 months.

SUMMARY:
Transitional psychiatry addresses the complex process through which individuals move from adolescence to adulthood, both in terms of developmental stage and mental healthcare systems. This transition includes the shift from pediatric to adult psychiatric services, as well as the evolution from vague or subclinical symptoms to established psychiatric disorders that may become chronic without early intervention.

Psychiatric disorders often emerge early in life: approximately 50% before age 15 and 75% before age 25. Early detection and intervention are therefore crucial to improving long-term mental health outcomes, functional independence, and social integration. However, current healthcare systems frequently fail to meet the needs of adolescents and young adults during this critical transition phase. Organizational discontinuities and clinical complexity lead to several risks:

* Difficulties in accessing appropriate psychiatric care for adolescents presenting with emerging symptoms,
* High rates of service disengagement for patients already receiving pediatric mental health care who do not successfully transition to adult services.

Studies have shown that nearly half (48%) of young people drop out of psychiatric follow-up for at least three months after reaching adulthood. This interruption increases the likelihood of relapse and involuntary psychiatric admissions. Despite numerous publications over the past decade emphasizing the need for dedicated transitional care models, services remain fragmented in many systems.

One of the largest recent studies in this area, the European MILESTONE longitudinal study, followed 763 patients (mean age 17.5) over two years in eight countries. It found that 11% of participants discontinued care entirely, 41% experienced discontinuity, and only 21% successfully transitioned to adult psychiatry. Continued care was more likely among patients with severe psychiatric disorders who had already accepted treatment. In contrast, those with mood disorders or poorly defined symptoms-despite being at high risk-were less likely to receive ongoing support.

Transitional psychiatry therefore aims to establish integrated practices and systems that ensure the continuity of mental healthcare for youth aged approximately 16 to 25. The main objectives of such services are to:

* Prevent care disruptions at the age of majority,
* Maintain appropriate and developmentally sensitive treatment for young adults,
* Promote patient autonomy in managing their care,
* Ensure coordination and collaboration between child/adolescent and adult psychiatric teams.

Despite growing recognition of these needs, no consensus exists in the literature regarding a fixed duration that defines a true care discontinuity, and practices vary significantly between regions and systems.

In this context, the Odyssée 3 project was launched in Nice, France, as a prospective epidemiological study focusing specifically on the real-life transition from child and adolescent psychiatry to adult psychiatry. The study targets a cohort of 17-year-olds who are currently receiving mental health care and will soon face the shift to adult services.

The project is part of the CNR Santé Mentale territorial initiative, supported by the Regional Health Agency (ARS 06). It is co-led by the University Department of Child and Adolescent Psychiatry (SUPEA) at Lenval Pediatric University Hospital and the Department of Psychiatry at the Nice University Hospital (CHU de Nice).

Odyssey 3 has three primary goals:

* To assess the care pathways and clinical outcomes of adolescents undergoing transition to adult psychiatry;
* To identify patient profiles, trajectories, and risk factors associated with successful or failed care continuity;
* To generate data that will inform the creation of a dedicated transitional psychiatry team and pathway in the Nice area.

Ultimately, this study aims to strengthen the healthcare system's ability to detect early warning signs, intervene proactively in emerging psychiatric conditions, and ensure that adolescents already engaged in care do not experience service discontinuities. Its findings will serve as a foundation for building a specialized, coordinated, and sustainable transitional psychiatry structure in Nice, aligned with best practices and international recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥17 and <18 years
* Living in the city of Nice
* Affiliated with the French national health insurance system
* French-speaking
* Signed informed consent from the patient and from one parent or legal guardian

Exclusion Criteria:

* Non

Ages: 17 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Group of 17-year-old patients living in Nice and receiving psychiatric care
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Annual prevalence of 17-year-old patients living in Nice who consulted hospital-based child and adolescent psychiatry services, calculated against the total number of 17-year-olds in the general population of Nice. | one year
  Annual prevalence is defined as the number of 17-year-old patients living in the city of Nice who consult hospital-based child and adolescent psychiatry services within a one-year period, divided by the total number of 17-year-olds in the general population of Nice. The calculation was performed using data from INSEE (French National Institute of Statistics and Economic Studies).

IPD SHARING:
Plan to Share IPD: Undecided